CLINICAL TRIAL: NCT01164007
Title: Phase II Study of Dacarbazine With the Anti-Vascular Endothelial Growth Factor Antibody (Bevacizumab) in Patients With Unresectable/Metastatic Melanoma
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Dacarbazine in Participants With Unresectable/Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18727; 2005-003416-30 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-16 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Dacarbazine

ARMS (1):
- Dacarbazine + Bevacizumab (Experimental): Participants with unresectable/metastatic melanoma not previously treated with chemotherapy for metastatic disease will receive dacarbazine and bevacizumab until disease progression, unacceptable toxicity, participant withdrawal, or physician decision to discontinue.
  Interventions: Drug: Bevacizumab; Drug: Dacarbazine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be given as 10 milligrams per kilogram (mg/kg) via intravenous (IV) infusion on Days 1 and 14 of each 28-day cycle.
  Other Names: Avastin
Drug: Dacarbazine — Dacarbazine will be given as 800 milligrams per square meter (mg/m^2) via IV infusion on Day 1 of each 28-day cycle.

SUMMARY:
This study will assess the preliminary anti-tumor activity and safety profile of a combination of bevacizumab and dacarbazine in participants with unresectable/metastatic melanoma not previously treated with chemotherapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cutaneous malignant melanoma
* Clinical evidence of metastatic disease and/or unresectable regional lymphatic disease and/or extensive in transit recurrent disease
* Measurable and/or evaluable lesions according to RECIST

Exclusion Criteria:

* Prior interferon alfa and/or cytokine therapy for metastatic disease
* Prior chemotherapy for metastatic disease
* Brain metastases
* Chronic daily treatment with high-dose aspirin (more than 325 milligrams per day)
* Other co-existing malignancies or malignancies diagnosed within the past 5 years with the exception of basal cell cancer or cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2012-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Istituto Europeo Di Oncologia, Milan, Lombardy, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Dacarbazine + Bevacizumab: Participants with unresectable/metastatic melanoma not previously treated with chemotherapy for metastatic disease received dacarbazine as 800 milligrams per square meter (mg/m^2) via intravenous (IV) infusion on Day 1 and bevacizumab as 10 milligrams per kilogram (mg/kg) via IV infusion on Days 1 and 14 of each 28-day cycle. Treatment continued until disease progression, unacceptable toxicity, participant withdrawal, or physician decision to discontinue.
Period: Overall Study
Arm/Group | Dacarbazine + Bevacizumab
Started | 40
Treated | 37
Completed | 0
Not Completed | 40
Not completed — Adverse Event | 5
Not completed — Progression of Disease | 30
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Medical Decision | 3

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who signed the Informed Consent Form (ICF) and received at least one dose of study medications.
Groups:
- Dacarbazine + Bevacizumab: Participants with unresectable/metastatic melanoma not previously treated with chemotherapy for metastatic disease received dacarbazine as 800 mg/m^2 via IV infusion on Day 1 and bevacizumab as 10 mg/kg via IV infusion on Days 1 and 14 of each 28-day cycle. Treatment continued until disease progression, unacceptable toxicity, participant withdrawal, or physician decision to discontinue.
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.16 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumor assessments were performed using RECIST. CR was defined as disappearance of all target and non-target lesions with normalization of tumor markers. PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to sum of LD at Baseline. Both were to be confirmed at a follow-up visit at least 4 weeks from the initial assessment of CR or PR. The percentage of participants with a best overall response of CR or PR during the study was reported.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: Intent-to-Treat (ITT) Population: All participants who signed the ICF, were assigned a study identifier, and received at least one dose of study medications.
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
percentage of participants | 18.92
Statistical Analysis 1: Comparison: Dacarbazine + Bevacizumab; The observed percentage of participants with CR or PR was compared with the expected proportion under the null hypothesis (0.10) and analyzed for statistical significance using a one-sample exact binomial test; Test type: Superiority or Other; p = 0.071, One-sample exact binomial test

2. Secondary Outcome: Percentage of Participants With Death or Disease Progression Following a Previous Assessment of CR or PR According to RECIST
Description: Tumor assessments were performed using RECIST. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). CR was defined as disappearance of all target and non-target lesions with normalization of tumor markers. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. The percentage of participants who died or demonstrated disease progression among those with a previous assessment of CR or PR was reported.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population. The "Number of Participants Analyzed" reflects the number of participants with a previous assessment of CR or PR.
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 7
percentage of participants | 57.14

3. Secondary Outcome: Duration of Response (DOR) With CR or PR According to RECIST
Description: Tumor assessments were performed using RECIST. DOR was defined as the time from first assessment of CR or PR to the time of death or disease progression, whichever occurred first. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). CR was defined as disappearance of all target and non-target lesions with normalization of tumor markers. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. DOR was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 7
months | 16.89 [5.77 to NA] — The upper limit could not be reached because of a high number of censored participants.

4. Secondary Outcome: Percentage of Participants With Death or Disease Progression Following a Previous Assessment of CR, PR, or Stable Disease (SD) According to RECIST
Description: Tumor assessments were performed using RECIST. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). CR was defined as disappearance of all target and non-target lesions with normalization of tumor markers. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for disease progression, using smallest sum of LD on study as reference. The percentage of participants who died or demonstrated disease progression among those with a previous assessment of CR, PR, or SD was reported.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population. The "Number of Participants Analyzed" reflects the number of participants with a previous assessment of CR, PR, or SD.
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 18
percentage of participants | 72.22

5. Secondary Outcome: DOR With CR, PR, or SD According to RECIST
Description: Tumor assessments were performed using RECIST. DOR was defined as the time from first assessment of CR, PR, or SD to the time of death or disease progression, whichever occurred first. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). CR was defined as disappearance of all target and non-target lesions with normalization of tumor markers. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for disease progression, using smallest sum of LD on study as reference. DOR was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 18
months | 12.52 [5.61 to 17.70]

6. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to RECIST
Description: Tumor assessments were performed using RECIST. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). The percentage of participants who died or demonstrated disease progression was reported.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
percentage of participants | 81.08

7. Secondary Outcome: Time to Progression (TTP) According to RECIST
Description: Tumor assessments were performed using RECIST. TTP was defined as the time from Baseline visit to time of death or disease progression, whichever occurred first. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). TTP was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
months | 5.48 [2.95 to 10.92]

8. Secondary Outcome: Percentage of Participants Who Discontinued Treatment
Description: The percentage of participants who discontinued treatment as a result of death, adverse event, disease progression, loss to follow-up, non-compliance, or consent withdrawal was reported. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s).
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
percentage of participants | 91.89

9. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from start of treatment to the time of treatment discontinuation as a result of death, adverse event, disease progression, loss to follow-up, non-compliance, or consent withdrawal was reported. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum on study or the appearance of new lesion(s). TTF was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
months | 3.05 [2.56 to 8.75]

10. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died from any cause was reported.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
percentage of participants | 81.08

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from Baseline visit to the time of death from any cause. OS was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Baseline up to approximately 6 years (assessed at Baseline, every 12 weeks on treatment, thereafter every 3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine + Bevacizumab
Number analyzed (Participants) | 37
months | 11.41 [6.46 to 25.11]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 6 years (assessed continuously on treatment)
Description: Safety Population
Arm/Group | Dacarbazine + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine + Bevacizumab (N=37)
Pyrexia (General disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Drug hypersensitivity (Immune system disorders) | 1
Influenza (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine + Bevacizumab (N=37)
Anaemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Conjunctivitis (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 10
General physical health deterioration (General disorders) | 2
Mucosal inflammation (General disorders) | 8
Pyrexia (General disorders) | 4
Influenza (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 4
Strangury (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.